CLINICAL TRIAL: NCT02339974
Title: Heterotopic Implantation Of the Edwards-Sapien Transcatheter Aortic Valve in the Inferior VEna Cava for the Treatment of Severe Tricuspid Regurgitation HOVER Trial
Brief Title: Heterotopic Implantation Of the Edwards-Sapien Transcatheter Aortic Valve in the Inferior VEna Cava for the Treatment of Severe Tricuspid Regurgitation (HOVER)
Acronym: HOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Brian O'Neill MD, Cardiologist, Temple University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G140131
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Severe Tricuspid Regurgitation (Experimental): This is a non-blinded (open label), non-randomized safety and feasibility study of the heterotopic implantation of the Edwards Sapien 3 valve.
  Interventions: Device: Heterotopic Implantation Of the Edwards-Sapien XT Transcatheter Valve in the Inferior VEna Cava

INTERVENTIONS:
Device: Heterotopic Implantation Of the Edwards-Sapien XT Transcatheter Valve in the Inferior VEna Cava

SUMMARY:
The goal of this study is to determine the short term safety (<30 days) and efficacy (6 months) of the heterotopic implantation of the Edwards-Sapien XT valve in the inferior vena cava for the treatment of severe tricuspid regurgitation in patients who are inoperable or at a very high surgical risk for tricuspid valve replacement.

DETAILED DESCRIPTION:
This is a prospective multi-center, non-blinded (open label), non-randomized safety and feasibility study of the heterotopic implantation of the Edwards-Sapien XT or S3 valve in the inferior vena cava for the treatment of severe tricuspid regurgitation in patients who are inoperable or at a very high surgical risk for tricuspid valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 21 years old.
2. The patient must have severe, symptomatic (ACC/AHA Stage D symptoms) tricuspid regurgitation (TR) as assessed by 2D echocardiogram with evidence of peripheral and central venous congestion (specifically lower extremity edema and abdominal ascites requiring diuretics.)
3. The patient must be evaluated by a "heart team" of physicians including an interventional cardiologist, cardiothoracic surgeon, heart failure specialist, and imaging specialist, and presented for review at a local multi-disciplinary conference. By consensus, the heart team must agree (and verify in the case review process) that valve implantation will likely benefit the patient.
4. The heart team must agree that medical factors preclude operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Also, other factors which may increase the patients perceived surgical risk for inclusion in the trial will be clearly delineated if they are present. These include, but are not limited to the following as defined by VARC 2: Frailty, Hostile chest, porcelain aorta, IMA or other critical conduit crossing the midline or adherent to the posterior table of sternum, severe right ventricular (RV) dysfunction. The surgeons' consultation notes shall specify the medical or anatomic factors leading to that conclusion. At least one of the cardiac surgeon assessors must have interviewed and examined the patient.
5. The study patient provides informed consent and agrees to comply with all required post-procedure follow-up visits, including annual visits up to 5 years.

Exclusion Criteria:

1. Heart Team assessment of operability (the heart team considers the patient to be a good surgical candidate).
2. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
3. Untreated, severe, left sided valvular heart disease including mitral regurgitation or stenosis, and aortic regurgitation or stenosis.
4. Mean pulmonary artery pressures ≥40mmHG and PVR >4 woods units as assessed by right heart catheterization.
5. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure. Examples of permanent implant would include any new heart valve. Implantation of a permanent pacemaker is excluded.
6. Patients with planned concomitant surgical or transcatheter ablation for Atrial Fibrillation.
7. Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mL).
8. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of screening evaluation.
9. Need for emergency surgery for any reason.
10. Left ventricular ejection fraction <40%.
11. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
12. Active upper GI bleeding within 3 months (90 days) prior to procedure.
13. A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
14. Recent CVA clinically confirmed (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 6 months (180 days) of the procedure.
15. Estimated life expectancy < 1 year from conditions other than TR.
16. Expectation that patient will not improve despite treatment of tricuspid regurgitation
17. Currently participating in another investigational cardiac device study or any other clinical trial, including drugs or biologics. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
18. Active bacterial endocarditis within 6 months (180 days) of procedure.
19. Patients with signs or symptoms of SVC syndrome, or hepatic cirrhosis not felt due to passive congestion from TR.

20: Subject unable to personally provide informed consent 21. FEV1<30% of predicted 22. Model for End State Liver Disease (MELD) score ≥21 (calculated per reference study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P O'Neill, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hosptial, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Tricuspid Regurgitation: This is a non-blinded (open label), non-randomized safety and feasibility study of the heterotopic implantation of the Edwards Sapien 3 valve.
  Heterotopic Implantation Of the Edwards-Sapien XT Transcatheter Valve in the Inferior VEna Cava
Period: Overall Study
Arm/Group | Severe Tricuspid Regurgitation
Started | 15
Completed | 7
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — Kansas City Cardiomyopathy Questionnaire (KCCQ) is a patient-reported measure of a patient's self-perceived health status scaled from 0 to 100. Scores are summarized in ranges to define patient health status: 0 to 24 is very poor to poor health, 25 to 49 is poor to fair health, 50 to 74 is fair to good health, 75 to 100 is good to excellent health. The baseline KCCQ is compared to KCCQ measures collected at follow-up to determine how an intervention affects a patient's self-perceived health status. This comparison is factored into Primary Outcome: Individual Patient Success.
  units on a scale | 52.4 (16.38)
6 Minute Walk Test [Mean (Standard Deviation); unit: Meters] — 6 Minute Walk Test (6MWT) measures exercise capacity by assessing the distance a person can walk in 6 minutes. When comparing baseline to follow-up 6MWT, further distance walked in 6 minutes corresponds to an increase in exercise capacity, shorter 6MWT distance corresponds to a decrease in exercise capacity. The baseline 6MWT is compared to 6MWT measures collected at follow-up to determine how an intervention affects patient exercise capacity. This comparison is factored into Primary Outcome: Individual Patient Success.
  Meters | 237.1 (138.14)

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: Procedural success will include both device success and no device/procedure related SAE's including: all death, all stroke, MI, new AKI grade 3, life threatening bleeding, major vascular complications (arterial or venous-requiring unplanned intervention), pericardial effusion or tamponade requiring drainage, SVC syndrome.
  Safety as defined by successful vascular access without unplanned major vascular complication as defined by VARC-2, delivery and retrieval of the transcatheter valve delivery system, correct position of both the vascular stent(s) and transcatheter valve in the IVC, a single valve placed within the IVC, and no need for additional surgery or re-intervention (including drainage of pericardial effusion) with the patient being alive at 30-days.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Percentage of Participants | 42.86 [9.90 to 81.59]

2. Primary Outcome: Individual Patient Success
Description: Individual patient success is defined by device success and the following: no re-hospitalizations for right sided heart failure or right sided heart failure equivalents including drainage of ascites or pleural effusions, new listing for heart transplant, VAD, or other mechanical support; improvement in one of three variables: KCCQ improvement>15 vs. baseline; 6MWT improvement> 70 meters vs. baseline; or VO2 peak improvement > 6% vs baseline..
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants | 2

3. Secondary Outcome: Lower Extremity Edema
Description: Measure of improvement in lower extremity (LE) edema measured by the Villalta Scale. The Villalta Scale is used to assess patients with lower extremity signs and symptoms of swelling, discoloration, or ulceration. The scale evaluates 5 patient reported items (pain, cramps, heaviness, paresthesia, pruritus) and 6 clinician-observed items (pretibial edema, skin induration, hyperpigmentation, pain during calf compression, venous ectasia, redness). Each item is graded on a four-point scale (0=none, 1=mild, 2=moderate, 3=severe). All points are added, resulting in an overall score from 0 to 33. The final Villalta score of 5-9 is mild disease, 10-14 is moderate, and ≥15 is severe disease. A 3.1 point reduction in this scale between time points is associated with improved quality of life.
Time Frame: 30 days, 6 months, 1 Year
Population: Incomplete data for these follow-up time frames.
Measure: Mean (Standard Deviation); unit: Villalta Scale Score
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Villalta Scale Score
  30 Days: number analyzed (Participants) | 6
  30 Days | 7.5 (4.23)
  6 Months: number analyzed (Participants) | 2
  6 Months | 9 (5.66)
  1 Year: number analyzed (Participants) | 3
  1 Year | 4.7 (5.51)

4. Secondary Outcome: Stroke and Transient Ischemic Attack (TIA)
Description: Occurrence of stroke or transient ischemic attack (TIA) by Valve Academic Research Consortium (VARC-2) criteria. VARC-2 diagnostic criteria defines stroke as a duration of a focal or global neurological deficit ≥ 24 hours; OR <24 hours if available neuroimaging documents a new hemorrhage or infarct; OR the neurological deficit results in death. VARC-2 diagnostic criteria defines TIA as a duration of a focal or global neurological deficit <24 hours, any variable neuroimaging does not demonstrate a new hemorrhage or infarct.
Time Frame: 30 days, 6 months, 1 year
Population: Incomplete data for these follow-up time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants
  30 Days: No Occurrence of Stroke or TIA | 6
  30 Days: Occurence of Stroke or TIA Occurrence | 1
  6 Months: number analyzed (Participants) | 4
  6 Months: No Occurrence of Stroke or TIA | 4
  6 Months: Occurence of Stroke or TIA Occurrence | 0
  1 Year: number analyzed (Participants) | 3
  1 Year: No Occurrence of Stroke or TIA | 1
  1 Year: Occurence of Stroke or TIA Occurrence | 2

5. Secondary Outcome: Mortality
Description: Mortality by Valve Academic Research Consortium (VARC-2) criteria. VARC-2 criteria separate All-cause mortality into 'Cardiovascular mortality' and 'Noncardiovascular mortality'. Cardiovascular mortality is defined as any of the following criteria: Death due to proximate cardiac cause (eg, myocardial infarction, cardiac tamponade, worsening heart failure); Death caused by noncoronary vascular conditions such as neurological events, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease; All procedure-related deaths, including those related to a complication of the procedure or treatment for a complication of the procedure; All valve-related deaths including structural or nonstructural valve dysfunction or other valve-related adverse events; Sudden or unwitnessed death; Death of unknown cause. Noncardiovascular mortality is defined as any death in which the primary cause of death is clearly related to another condition (eg, trauma, cancer, suicide)
Time Frame: 30 days, 6 months, 1 year
Population: Incomplete data for these follow-up time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants
  30 Days: No Occurrence of Death | 6
  30 Days: Occurrence of Death | 1
  6 Months: number analyzed (Participants) | 4
  6 Months: No Occurrence of Death | 2
  6 Months: Occurrence of Death | 2
  1 Year: number analyzed (Participants) | 3
  1 Year: No Occurrence of Death | 1
  1 Year: Occurrence of Death | 2

6. Secondary Outcome: Myocardial Infarction
Description: Myocardial Infarction (MI) by Valve Academic Research Consortium (VARC-2) criteria. VARC-2 defines MI as either periprocedural MI (new ischemic symptoms or signs AND elevated cardiac biomarkers within 72 hours after the index procedure), or spontaneous MI (>72hours after the index procedure, any 1 of the following: detection of rise and/or fall of cardiac biomarkers with at least 1 value above the 99th percentile, together with the evidence of myocardial ischemia with either symptoms of ischemia, ECG changes indicative of new ischemia, new pathological Q-waves in at least two contiguous leads, or imaging evidence of a new loss of viable myocardium or new wall motion abnormality; Sudden, unexpected cardiac death involving cardiac arrest, accompanied by new ST elevation or new LBBB, and/or evidence of fresh thrombus by coronary angiogram or at autopsy, or at a time before the appearance of cardiac biomarker in the blood; or Pathological findings of an acute MI).
Time Frame: 30 days, 6 months, 1 Year
Population: Incomplete data for these follow-up time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants
  30 Days: No Occurrence of MI | 7
  30 Days: Occurrence of MI | 0
  6 Months: number analyzed (Participants) | 4
  6 Months: No Occurrence of MI | 4
  6 Months: Occurrence of MI | 0
  1 Year: number analyzed (Participants) | 3
  1 Year: No Occurrence of MI | 3
  1 Year: Occurrence of MI | 0

7. Secondary Outcome: Acute Kidney Injury
Description: Occurrence of Acute Kidney Injury (AKI) by Valve Academic Research Consortium (VARC-2) criteria. VARC-2 criteria defines AKI as any of the following: [Stage 1] Increase in serum creatinine to 150-199% OR Urine output <0.5mL/kg/h for >6 but <12hours; [Stage 2] Increase in serum creatinine to 200-299% OR Urine output <0.5 mL/kg/h for >6 but <12hours; or [Stage 3] Increase in serum creatinine to ≥300% OR Urine output <0.3mL/kg/h for ≥24hours OR Anuria for ≥12hours.
Time Frame: 30 days, 6 months, 1 Year
Population: Incomplete data for these follow-up time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants
  30 Days: No Occurrence of Acute Kidney Injury | 5
  30 Days: Occurrence of Acute Kidney Injury | 2
  6 Months: number analyzed (Participants) | 4
  6 Months: No Occurrence of Acute Kidney Injury | 4
  6 Months: Occurrence of Acute Kidney Injury | 0
  1 Year: number analyzed (Participants) | 3
  1 Year: No Occurrence of Acute Kidney Injury | 2
  1 Year: Occurrence of Acute Kidney Injury | 1

8. Secondary Outcome: Major Vascular Complications
Description: Major Vascular Complications by Valve Academic Research Consortium (VARC-2) criteria. VARC-2 defines major vascular complications as: any aortic dissection aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudoaneurysm; Access site or access-related vascular injury leading to death, life threatening or major bleeding, visceral ischemia, or neurological impairment; Distal embolization from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage; The use of unplanned endovascular or surgical intervention associated with death, major bleeding, visceral ischemia or neurological impairment; Any new ipsilateral lower extremity ischemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram; surgery for access site-related nerve injury; or Permanent access site-related nerve injury.
Time Frame: 30 days, 6 months, 1 Year
Population: Incomplete data for these follow-up time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Tricuspid Regurgitation
Number analyzed (Participants) | 7
Participants
  30 Days: No Occurrence of Major Vascular Complication | 6
  30 Days: Occurrence of Major Vascular Complication | 1
  6 Months: number analyzed (Participants) | 4
  6 Months: No Occurrence of Major Vascular Complication | 4
  6 Months: Occurrence of Major Vascular Complication | 0
  1 Year: number analyzed (Participants) | 3
  1 Year: No Occurrence of Major Vascular Complication | 1
  1 Year: Occurrence of Major Vascular Complication | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Severe Tricuspid Regurgitation
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Tricuspid Regurgitation (N=7)
Stroke and TIA (Nervous system disorders) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3)
Major vascular complications (Vascular disorders) | 3 (3)
Lower Extremity Edema (Cardiac disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Tricuspid Regurgitation (N=7)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an early feasibility study. The study did not achieve its intended enrollment of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT02339974/Prot_SAP_ICF_000.pdf